CLINICAL TRIAL: NCT00559533
Title: A Multi-center, Open-label, Phase I Study of Single Agent R7112 Administered Orally in Patients With Advanced Malignancies, Except All Forms of Leukaemia
Brief Title: A Study of RO5045337 [RG7112] in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO21280
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RO5045337

INTERVENTIONS:
Drug: RO5045337 — Administered po at escalating doses (with a starting dose of 20mg/m2/day) (5-10 cohorts)

SUMMARY:
This study will determine the maximum tolerated dose and the optimal associated 4 weekly dosing schedule of RO5045337, administered as monotherapy in patients with advanced solid tumors. A first cohort of patients will receive the starting dose of 20mg/m2/day, once daily for 10 days in each 28 day cycle. Subsequent cohorts of patients will receive dose escalations, and possible changes in dosing schedule, based on tolerability and pharmacokinetic knowledge gained from prior treatment cohorts. The anticipated time on study treatment is until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* solid tumor malignancies;
* failed prior therapies, or no standard therapy available;
* ECOG performance status of 0-2.

Exclusion Criteria:

* patients receiving any other agent or therapy to treat their malignancy;
* pre-existing gastrointestinal disorders which may interfere with absorption of drugs;
* clinically significant cardiovascular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
MTD and associated dose schedule | Every 28 days

SECONDARY OUTCOMES:
Clinical response | Event driven
Dose-limiting toxicities. | Throughout study
Pharmacokinetic profile | Throughout study
Comparison safety and tolerability of daily versus twice daily dosing regimens | approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (5):
  - Aurora, Colorado
  - Boston, Massachusetts
  - New York, New York
  - Houston, Texas
  - San Antonio, Texas
- France (2):
  - Bordeaux
  - Lyon